CLINICAL TRIAL: NCT03050684
Title: Does Vaginal Washing Before Inserting Dinoprostone Affect the Success Rate of the Labour Induction?
Brief Title: Does Vaginal Washing Affect the Success Rate of the Labour Induction?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Çiğdem Yayla Abide, Ob&Gyn Specialist, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Screening
Other Study IDs: 2016-162
Record Dates: First submitted 2017-01-21; First posted 2017-02-13 (Actual); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Labor Induction; Dinoprostone Vaginal Insert; Vaginal Infection; Effect Increased
MeSH Terms: conditions — Vaginitis | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- vaginal lavage group (Active Comparator): We will make vaginal lavage with steril %0.9 NaCl serum ( 20cc) before inserting dinoprostone (Propess ®) 10 mg vaginal ovule
  Interventions: Procedure: vaginal lavage group
- Control group (Placebo Comparator): We will insert dinoprostone (Propess ®) vaginal ovule without vaginal lavage.
  Interventions: Procedure: Control Group

INTERVENTIONS:
Procedure: vaginal lavage group — vaginal washing will be applied with steril %0.9 NaCl serum (20cc) before intravaginal PGE2 insertion.
  Arms: vaginal lavage group
Procedure: Control Group — vaginal washing will be not applied with steril %0.9 NaCl serum (20cc) before intravaginal PGE2 insertion.
  Arms: Control group

SUMMARY:
Investigators will use dinoprostone(Propess TM) for cervix ripening and labor induction in term pregnant women.Vaginal pH base is achieved with the effect of hormones in pregnancy and associated with this, vaginal infections rates increase. With the vaginal application of Propess, the preparate remains in the vagina for a long time, with controlled release,creating a film layer against bacteria and especially fungal infections and it was thought that this could be a reason for unsuccessful birth induction by preventing release of this ovule.

The aim of this study is to observe whether or not the rate of caesareans with the indication of unsuccessful induction was reduced in patients by reducing the density of vaginal bacteria and fungi with vaginal lavage and thereby increasing the effect of the drug and decreasing the rate of unsuccessful inductions.

DETAILED DESCRIPTION:
The study will include patients meeting the study criteria monitored in the delivery .

Verbal and written informed consent will be obtained from all patients before starting the study. The patients will be randomised to 2 groups. In one group, vaginal lavage (the vagina will first be washed with saline in a 20cc injector) will be applied then Propess will be used and in the other group Propess will be used without any lavage.

It is planned to include 70 patients in each group.

ELIGIBILITY:
Inclusion Criteria:

* Patients with singleton pregnancies
* Term gestational week (defined as>37 weeks),
* Fetal cephalic presentation
* Participiants with with intact amniotic membrane
* Reactive fetal heart rate
* Cervical Modified Bishop's score <5

Exclusion Criteria:

* Patients with with multipl pregnancies
* Participiants with malpresentation anomalies
* Participiants with nonreassurring fetal heart rate
* Participiants with more than three contractions in 10 minutes
* Participiants with contrandications for using prostaglandins
* Participiants with fetal anomaly
* Participiants with fetal demise
* Participiants with emercency delivery indications,
* Participiants with previous cesarean delivery or have other uterine surgery
* Participiants with cephalopelvic disproportion

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2017-02-20 (Actual); Primary Completion 2017-12-10 (Actual); Study Completion 2017-12-20 (Actual)

PRIMARY OUTCOMES:
Succesful cervical repining which allows succesful vaginal delivery | 12 Months
  Cervical ripening is defined cervical Bishop score >5 the indication of unsuccessful induction

CONTACTS AND LOCATIONS:
Overall Officials: İlter Yenidede, MD, Principal Investigator — Zeynep Kamil Maternity and Children Hospital; Çetin Kılıççı, Principal Investigator — Zeynep Kamil Maternity and Children Hospital
Locations (1):
- Zeynep Kamil Maternity and Children Hospital, Istanbul, Turkey (Türkiye)